CLINICAL TRIAL: NCT04458909
Title: An Open-Label, Phase III Study of Platinum-Gemcitabine With or Without Nivolumab in the First-Line Treatment of Recurrent or Metastatic Nasopharyngeal Carcinoma
Brief Title: Testing the Addition of an Anti-cancer Immune Therapy Drug (Nivolumab) to the Usual Chemotherapy Treatment (Cisplatin or Carboplatin With Gemcitabine) for Recurrent or Metastatic Nasopharyngeal Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: External information
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-04581; NCI-2020-04581 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-HN007 (Other: NRG Oncology); NRG-HN007 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Nasopharyngeal Carcinoma; Metastatic Nasopharyngeal Keratinizing Squamous Cell Carcinoma; Metastatic Nasopharyngeal Nonkeratinizing Carcinoma; Metastatic Nasopharyngeal Undifferentiated Carcinoma; Nasopharyngeal Nonkeratinizing Carcinoma; Recurrent Nasopharyngeal Carcinoma; Recurrent Nasopharyngeal Keratinizing Squamous Cell Carcinoma; Recurrent Nasopharyngeal Undifferentiated Carcinoma; Stage IV Nasopharyngeal Carcinoma AJCC v8; Stage IVA Nasopharyngeal Carcinoma AJCC v8; Stage IVB Nasopharyngeal Carcinoma AJCC v8
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Gemcitabine; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (nivolumab, gemcitabine, cisplatin / carboplatin) (Experimental): Patients receive nivolumab IV over 30 minutes on day 1, gemcitabine IV over 30 minutes on days 1 and 8, and cisplatin IV over 30-60 minutes or carboplatin IV over 30-60 minutes on day 1. Treatment repeats every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity. After 4 weeks, patients then receive nivolumab IV over 30 minutes on day 1. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Drug: Gemcitabine; Biological: Nivolumab; Other: Questionnaire Administration
- Arm II (gemcitabine, cisplatin / carboplatin) (Active Comparator): Patients receive gemcitabine and cisplatin or carboplatin as in Arm I.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Drug: Gemcitabine; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Gemcitabine — Given IV
  Other Names: dFdC; dFdCyd; Difluorodeoxycytidine
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BMS-936558; CMAB819; MDX-1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar CMAB819; ONO-4538; Opdivo
  Arms: Arm I (nivolumab, gemcitabine, cisplatin / carboplatin)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase III trial compares the effect of adding nivolumab to the usual chemotherapy (cisplatin or carboplatin with gemcitabine) versus standard chemotherapy alone in treating patients with nasopharyngeal cancer that has come back (recurrent) or spread to other places in the body (metastatic). Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Chemotherapy drugs, such as cisplatin, carboplatin, and gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving nivolumab with the usual chemotherapy may work better than the standard chemotherapy alone in treating patients with nasopharyngeal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if adding nivolumab to platinum-gemcitabine as first-line treatment improves overall survival (OS) for patients with recurrent and/or metastatic nasopharyngeal carcinoma (NPC).

SECONDARY OBJECTIVES:

I. To compare patterns of failure (local-regional relapse and distant metastasis) between treatment arms.

II. To determine if adding nivolumab to platinum-gemcitabine as first-line treatment improves the objective tumor response based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

III. To determine if adding nivolumab to platinum-gemcitabine as first-line treatment improves progression free survival (PFS) for patients with recurrent and/or metastatic NPC.

IV. To evaluate the toxicity based on the Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0.

V. To characterize patient-reported symptomatic toxicities measured by Patient-Reported Outcomes (PRO)-CTCAE.

VI. To assess the quality of life (QOL), as measured by the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-Core (C)30, between the two arms (primary PRO).

VII. To assess fatigue, as measured by Multidimensional Fatigue Inventory (MFI-20), between the two arms (secondary PRO).

VIII. To determine if a subset of patients based on an optimal cutoff point of Programmed Death Receptor Ligand-1 (PD-L1) Combined Positive Score (CPS)/Tumor Proportion Score (TPS) is more likely to benefit in terms of PFS from adding nivolumab to platinum-gemcitabine as first-line treatment.

EXPLORATORY OBJECTIVES:

I. To determine if a subset of patients based on an optimal cutoff point of PD-L1 CPS/TPS is more likely to benefit in terms of overall survival (OS) from adding nivolumab to platinum-gemcitabine as first-line treatment.

II. To determine changes in QOL as measured by EORTC QLQ-C30 and in fatigue as measured by MFI-20, between and within arms over time (exploratory PRO).

III. To collect blood and tissue specimens for future translational research.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive nivolumab intravenously (IV) over 30 minutes on day 1, gemcitabine IV over 30 minutes on days 1 and 8, and cisplatin IV over 30-60 minutes or carboplatin IV over 30-60 minutes on day 1. Treatment repeats every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity. After 4 weeks, patients then receive nivolumab IV over 30 minutes on day 1. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive gemcitabine and cisplatin or carboplatin as in Arm I.

After completion of study treatment, patients are followed up every 4 months for 2 years, every 6 months for 3 years, and then annually.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) proven diagnosis of NPC that has recurred at locoregional and/or distant sites. For locoregional recurrence, the disease must not be amenable to potentially curative surgery or re-irradiation. The following histological types are accepted: (a) Keratinizing - squamous cell carcinoma; (b) Non-keratinizing - undifferentiated or poorly differentiated
* Measurable disease by the RECIST 1.1 criteria. Lesion(s) that have been irradiated previously can be counted as measurable as long as radiological progression has been demonstrated prior to enrollment
* History/physical examination by a medical oncologist or clinical oncologist within 14 days prior to registration
* Zubrod/Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 within 14 days prior to registration
* Contrast enhanced magnetic resonance imaging (MRI) or computed tomography (CT) of the nasopharynx and neck within 30 days prior to registration
* Contrast enhanced CT scan of the chest, abdomen, and pelvis within 30 days prior to registration
* Absolute neutrophil count (ANC) >= 1500 cells/mm^3 (within 14 days prior to registration)
* Platelets >= 100,000 cells/mm^3 (within 14 days prior to registration)
* Hemoglobin >= 9.0 g/dL (transfusion is accepted. Erythropoietin dependency not accepted) (within 14 days prior to registration)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) OR direct bilirubin =< ULN for patients with total bilirubin levels > 1.5 x ULN. Patients with known Gilbert's syndrome are not excluded (within 14 days prior to registration)
* Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN (=< 3 x ULN for patients with liver metastases) (within 14 days prior to registration)
* Serum creatinine =< 1.5 x ULN OR calculated creatinine clearance (CrCl) based on Cockcroft-Gault equation >= 30 mL/min for patients with serum creatinine levels > 1.5 x ULN. In this protocol, cisplatin or carboplatin may be used at the discretion of the investigator - except for patients with CrCl between 30-50 mL/min, for whom carboplatin should be used instead of cisplatin (within 14 days prior to registration)
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable, and patients must be receiving anti-viral therapy at enrollment. Patients must agree to continue anti-viral therapy throughout the study period as directed by their treating physicians

  * Known positive test for hepatitis B virus surface antigen (HBsAg) indicating acute or chronic infection would make the patient ineligible unless the viral load becomes undetectable on anti-viral therapy
  * Patients who are immune to hepatitis B (anti-Hepatitis B surface antibody positive) are eligible (i.e., patients immunized against hepatitis B)
  * In some centers, hepatitis B core antibody (anti-HBc) is done routinely before chemotherapy for some cancer patients. This is because patients who are HBsAg-negative but positive for anti-HBc should have undetectable HBV viral load at enrollment and receive prophylactic anti-viral therapy throughout the study (American Society of Clinical Oncology 2015 guideline, Hwang 2015). In this protocol, anti-HBc should be performed based on institutional standards
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment they are eligible if they have an undetectable HCV viral load

  * Note: Known positive test for hepatitis C virus ribonucleic acid (HCV RNA) indicating acute or chronic infection would make the patient ineligible unless the viral load becomes undetectable on suppressive therapy
* For women of childbearing potential (WOCBP), negative serum or urine pregnancy test within 14 days prior to registration. For WOCBP randomized to Arm 1, an additional negative serum or urine pregnancy is required within 24 hours prior to starting nivolumab treatment

  * Women of childbearing potential (WOCBP) is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes
* Women of childbearing potential (WOCBP) and men who are sexually active with WOCBP must be willing to use an adequate method of contraception. Women must use an effective oral contraception and the male partner must use condom) during and after treatment
* The patient or a legally authorized representative must provide written informed consent prior to study entry

Exclusion Criteria:

* Diagnosed with another invasive malignancy (except non-melanomatous skin cancer) unless disease free for more than 3 years. Note: Patients with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) who have undergone potentially curative therapy are not excluded
* Any prior systemic anti-cancer agents (including chemotherapy and investigational agents) for the purpose of treating locoregional and/or distant recurrence of NPC
* Patients who have received neoadjuvant (induction) and/or adjuvant chemotherapy for primary NPC with chemotherapy (any drug regimens including those containing platinum and/or gemcitabine) at or within 6 months prior to registration are excluded (counting from the last day of the chemotherapy for the primary NPC, prior to enrolling into the current study). The following subgroups of patients are NOT excluded:

  * Patients who have received neoadjuvant (induction) and/or adjuvant chemotherapy for primary (non-metastatic/non-recurrent) NPC more than 6 months prior to registration, counting from the last day of the chemoradiotherapy for the primary NPC, prior to enrolling into the current study
  * For prior RT with radical intent: Patients who have prior radiotherapy (RT) to the primary and locoregional disease (i.e. non-recurrent disease) with or without concurrent cisplatin or carboplatin monotherapy are not excluded as long as they have not received any neoadjuvant/adjuvant chemotherapy within 6 months prior to registration (counting from the last day of the chemotherapy), and that the last RT fraction (with radical intent) has been given more than 3 months prior to registration
  * For RT with palliative intent: Prior radiotherapy (RT) at or within 30 days prior to registration, this includes RT given with palliative intent (with or without concurrent cisplatin or carboplatin alone) to recurrent/ metastatic sites in patients with recurrent/metastatic NPC. The re-irradiated sites must not be the only sites of measurable recurrent disease
  * Prior chemotherapy for cancers other than NPC is allowed as long as the last course of chemotherapy was administered more than 3 years prior to registration and the patient has remained disease-free for more than 3 years
* Prior therapy for any indication, with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g. CTLA-4, OX-40, CD137)
* History of severe (grade 3-4) hypersensitivity reaction to any monoclonal antibody including nivolumab and/or any of its excipients
* Severe, active co-morbidity defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
  * Myocardial infarction within the last 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days of registration
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
  * History of (non-infectious) pneumonitis that required steroids or has current pneumonitis requiring steroids and/or immunosuppressive therapy
  * History of active TB (Bacillus tuberculosis, not known to be multi-drug resistant) as defined by the need to receive systemic treatment within the last 2 years or any known history of multi-drug resistant TB. Note: Patients who had a distant history of treated TB (not known to be multi-drug resistant) at 5 or more years from enrollment and have no current symptoms suggestive of active TB, are not excluded from this study. Note: Testing for prior exposure to TB is not required in this study since TB is endemic in parts of Asia
  * Prior solid organ transplant or bone marrow transplant
  * History of active primary immunodeficiency including, but not limited to acquired immune deficiency syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition; Note: Human immunodeficient virus (HIV) testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatment involved in this protocol may be immunosuppressive
  * Condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone or equivalents) or other immunosuppressive medications within 14 days of registration. Inhaled or topical steroids and adrenal replacement doses < 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. Steroid premedication for the prophylaxis of CT contrast-related allergies is allowed. The use of dexamethasone as an anti-emetic premedication prior to chemotherapy is also allowed
  * Active autoimmune disease requiring systemic treatment (i.e. disease modifying agents, corticosteroids, or immunosuppressive drugs) within the past 2 years. These include but are not limited to patients with a history of immune-related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis; systemic autoimmune disease such as systemic lupus erythematosus (SLE), rheumatoid arthritis, connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome should be excluded because of the risk of recurrence or exacerbation of disease
  * Note: Patients are permitted to enroll if they have vitiligo; type I diabetes mellitus; hypothyroidism, pituitary or adrenal insufficiency requiring only hormone replacement; psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger (precipitating event)
* Patients who are pregnant or breastfeeding and unwilling to discontinue breastfeeding
* Known history of grade 3-4 allergic reaction and/or hepatic toxicity to cisplatin, carboplatin, or gemcitabine

  * Note: For patients with known history of grade 3-4 renal toxicity to cisplatin or known history of clinically significant hearing loss (grade 2 or above) attributed to cisplatin, or other intolerances to cisplatin that are of clinical significance, carboplatin can be used in this study and therefore these patients are NOT excluded from enrollment
* Known central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with base of skull involvement by NPC are not excluded unless their disease is directly invading the brain parenchyma and is associated with clinical symptoms (headaches, nausea and vomiting, neurological abnormalities on physical examination) and/or cerebral edema on radiological imaging
* Patients who have received a live vaccine within 30 days prior to the first dose of study treatment. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster, yellow fever, rabies, Bacillus Calmette-Guerin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist) are live attenuated vaccines and are not allowed
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brigette B Ma, Principal Investigator — NRG Oncology
Locations (325):
- United States (322):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Epic Care-Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Epic Care Cyberknife Center, Walnut Creek, California
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Saint Anthony's Health, Alton, Illinois
  - Rush - Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Reid Health, Richmond, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Mission Cancer and Blood - Laurel, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - Trinity Regional Medical Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Our Lady of the Lake Physicians Group - Medical Oncology, Baton Rouge, Louisiana
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China Township, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Academic Hematology Oncology Specialists, Grosse Pointe Woods, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Michigan Breast Specialists-Grosse Pointe Woods, Grosse Pointe Woods, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Medical Campus, Macomb, Michigan
  - Michigan Breast Specialists-Macomb Township, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - 21st Century Oncology-Pontiac, Pontiac, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Great Lakes Cancer Management Specialists-Rochester Hills, Rochester Hills, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Ascension Saint Joseph Hospital, Tawas City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Michigan Breast Specialists-Warren, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford South University Medical Center, Fargo, North Dakota
  - Southpointe-Sanford Medical Center Fargo, Fargo, North Dakota
  - Sanford Medical Center Fargo, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Saint Elizabeth Boardman Hospital, Boardman, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC-Miami Valley Hospital North, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Joseph Warren Hospital, Warren, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Saint Elizabeth Youngstown Hospital, Youngstown, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada
- Chinese University of Hong Kong-Prince of Wales Hospital, Shatin, Hong Kong, China
- National Cancer Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm II (Gemcitabine, Cisplatin / Carboplatin): Gemcitabine and cisplatin or carboplatin as in Arm I.
Period: Overall Study
Arm/Group | Arm I (Nivolumab, Gemcitabine, Cisplatin / Carboplatin) | Arm II (Gemcitabine, Cisplatin / Carboplatin)
Started | 11 | 4
Started Protocol Treatment | 11 | 4
Completed | 11 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Nivolumab, Gemcitabine, Cisplatin / Carboplatin) | Arm II (Gemcitabine, Cisplatin / Carboplatin) | Total
Number analyzed (Participants) | 11 | 4 | 15
Age, Customized [Count of Participants; unit: Participants]
  ≤ 49 years | 3 | 2 | 5
  50 - 59 years | 1 | 2 | 3
  60 - 69 years | 5 | 0 | 5
  ≥ 70 years | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 10 | 1 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 10 | 3 | 13
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 3 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 1 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Failure is death from any cause. Survival rates were to be estimated using the Kaplan-Meier method and arms were to be compared using a log-rank test. Analysis was to occur after 200 deaths have been reported. Given the small number of participants due to early study closure, only the number of patients last reported to be alive at time of study termination is reported.
Time Frame: Baseline to the date of death or last follow-up. Maximum follow-up time was 2.3 years.
Population: Randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Nivolumab, Gemcitabine, Cisplatin / Carboplatin) | Arm II (Gemcitabine, Cisplatin / Carboplatin)
Number analyzed (Participants) | 11 | 4
Participants | 8 | 4

2. Secondary Outcome: Locoregional Failure
Description: Locoregional failure is defined as first evidence of local or regional progression, death due to study cancer without documented progression, or death due to unknown causes without documented progression; distant metastasis and deaths from other causes were considered competing risks. Progressive disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 is defined as at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance or recurrence of any locoregional lesions is also considered progression. Failure rates were to be estimated using the cumulative incidence method and arms were to be compared using the cause-specific log-rank test. Analysis was to occur after 200 deaths. Given the small number of participants due to early study closure, only the number of patients with locoregional failure is reported.
Time Frame: Baseline to the date of failure or last known follow-up. Maximum follow-up time was 2.3 years.
Population: Randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Nivolumab, Gemcitabine, Cisplatin / Carboplatin) | Arm II (Gemcitabine, Cisplatin / Carboplatin)
Number analyzed (Participants) | 11 | 4
Participants | 6 | 0

3. Secondary Outcome: Distant Metastases
Description: Distant failure is defined as first evidence of distant metastasis; locoregional failure and all deaths were to be considered competing risks. Distant failure rates were to be estimated using the cumulative incidence method and arms were to be compared using the cause-specific log-rank test. Analysis was to occur after 200 deaths. Given the small number of participants due to early study closure, only the number of patients with distant failure is reported.
Time Frame: Randomization to the date of failure or last known follow-up. Maximum follow-up time was 2.3 years.
Population: Randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Nivolumab, Gemcitabine, Cisplatin / Carboplatin) | Arm II (Gemcitabine, Cisplatin / Carboplatin)
Number analyzed (Participants) | 11 | 4
Participants | 2 | 1

4. Secondary Outcome: Progression-free Survival (PFS)
Description: Failure is defined as local, regional, or distant disease progression, or death from any cause. Progressive disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 is defined as at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance or recurrence of any lesions is also considered progression. Failure rates were to be estimated using the Kaplan-Meier method and arms were to be compared using the log-rank test. Analysis was to occur after 200 deaths. Given the small number of participants due to early study closure, only the number of patients alive without progression is reported.
Time Frame: Baseline to the date of failure or last known follow-up. Maximum follow-up time was 2.3 years.
Population: Randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Nivolumab, Gemcitabine, Cisplatin / Carboplatin) | Arm II (Gemcitabine, Cisplatin / Carboplatin)
Number analyzed (Participants) | 11 | 4
Participants | 3 | 3

5. Secondary Outcome: Number of Participants With Complete or Partial Response (Objective Response Rate) Through the End of Cycle 6 Determined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Description: CT/MRI of nasopharynx and neck or chest CT at baseline and through the end of cycle 6 are compared to determine tumor response.
  Per RECIST 1.1:
  * Complete response:
    * Disappearance of all lesions and pathologic lymph nodes
  * Partial response:
    * 30% decrease sum of the longest diameters
      * No new lesions
      * No progression of non-target lesions
Time Frame: Baseline through end of cycle 6 (each cycle is 21 days)
Population: Randomized participants with scans at baseline and end of cycle 6
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Nivolumab, Gemcitabine, Cisplatin / Carboplatin) | Arm II (Gemcitabine, Cisplatin / Carboplatin)
Number analyzed (Participants) | 11 | 4
Participants | 4 | 0

6. Secondary Outcome: Number of Participants With Grade 3 or Higher Adverse Events (AEs)
Description: Common Terminology Criteria for Adverse Events (CTCAE) version 5 grades adverse event severity from 1=mild to 5=death. Summary data is provided in this outcome measure; see Adverse Events Module for specific adverse event data. Counts of participants with any grade 3 or higher adverse event are reported. Adverse events of any attribution are included.
Time Frame: Baseline to the date of last follow-up. Maximum follow-up time was 2.3 years.
Population: Randomized participants
Measure: Count of Participants; unit: Participants
Groups:
- Arm I (Nivolumab, Gemcitabine, Cisplatin / Carboplatin): Six cycles (3 weeks each):
  * Nivolumab 360 mg fixed dose IV over 30 minutes on day 1.
  * Cisplatin 80 mg/m^2 IV over 30-60 minutes or carboplatin AUC of 5 on day 1.
  * Gemcitabine 1000 mg/m^2 IV over 30 minutes on days 1 and 8.
  Followed by maintenance therapy for up to 24 cycles (4 weeks each):
  * Nivolumab 480 mg fixed dose IV over 30 minutes on day 1.
Arm/Group | Arm I (Nivolumab, Gemcitabine, Cisplatin / Carboplatin) | Arm II (Gemcitabine, Cisplatin / Carboplatin)
Number analyzed (Participants) | 11 | 4
Participants | 10 | 2

7. Secondary Outcome: Number of Participants With Patient Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) Severity Score ≥ 3 (or Present) at Baseline
Description: PRO-CTCAE is a patient-reported outcome (PRO) measurement system developed to evaluate symptomatic toxicity in patients on cancer clinical trials. This study collects PRO-CTCAE data on sixteen symptomatic adverse events (AEs), asking about experience over the last seven days. Worst severity of the given symptom was collected for 14 items (0=none, 1=mild, 2=moderate, 3=severe, and 4=very severe). Any presence of the symptom was collected for 2 items (present/absent). For each symptom, the row label indicates whether severity score ≥ 3 or presence is reported.
Time Frame: Baseline
Population: Randomized participants with any PRO-CTCAE data
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Nivolumab, Gemcitabine, Cisplatin / Carboplatin) | Arm II (Gemcitabine, Cisplatin / Carboplatin)
Number analyzed (Participants) | 9 | 3
Participants
  Dry mouth (severity grade 3+) | 1 | 1
  Difficulty swallowing (severity grade 3+) | 1 | 0
  Voice quality changes (presence) | 2 | 0
  Mouth/throat sore (severity grade 3+) | 0 | 0
  Taste changes (severity grade 3+) | 0 | 0
  Abdominal pain (severity grade 3+) | 0 | 0
  Heart palpitations (severity grade 3+) | 0 | 1
  Rash (presence) | 1 | 0
  Itching (severity grade 3+) | 0 | 0
  Numbness & tingling (severity grade 3+ | 0 | 0
  Blurred vision (severity grade 3+) | 0 | 0
  Ringing in ears (severity grade 3+) | 0 | 0
  Concentration (severity grade 3+) | 0 | 0
  Memory (severity grade 3+) | 1 | 0
  Headache (severity grade 3+) | 0 | 0
  Sad (severity grade 3+) | 0 | 0

8. Secondary Outcome: Number of Participants With Patient Reported Outcomes-Common Terminology Criteria for Adverse Events (PRO-CTCAE) Severity Score ≥ 3 (or Present) at Cycle 6
Description: as for outcome 7
Time Frame: End of cycle 6 (each cycle is 21 days for the first six cycles)
Population: Randomized participants with any PRO-CTCAE data
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Nivolumab, Gemcitabine, Cisplatin / Carboplatin) | Arm II (Gemcitabine, Cisplatin / Carboplatin)
Number analyzed (Participants) | 9 | 3
Participants
  Dry mouth (severity grade 3+) | 1 | 0
  Difficulty swallowing (severity grade 3+) | 0 | 0
  Voice quality changes (presence) | 1 | 0
  Mouth/throat sore (severity grade 3+) | 1 | 0
  Taste changes (severity grade 3+) | 0 | 0
  Abdominal pain (severity grade 3+) | 0 | 0
  Heart palpitations (severity grade 3+) | 0 | 0
  Rash (presence) | 1 | 0
  Itching (severity grade 3+) | 0 | 0
  Numbness & tingling (severity grade 3+ | 0 | 0
  Blurred vision (severity grade 3+) | 0 | 0
  Ringing in ears (severity grade 3+) | 0 | 0
  Concentration (severity grade 3+) | 0 | 0
  Memory (severity grade 3+) | 1 | 0
  Headache (severity grade 3+) | 0 | 0
  Sad (severity grade 3+) | 0 | 0

9. Secondary Outcome: Global Heath Status (GHS) Score of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30)
Description: Global Health Status is calculated from two questions on the EORTC QLQ-C30. The question responses range from 1 "very poor" to 7 "excellent" such that a higher response indicates better quality of life (QOL). The mean of these responses is linearly transformed to a range of 0 (worst) to 100 (best).
Time Frame: End of cycle 6 (each cycle is 21 days)
Population: Randomized participants with cycle 6 data
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Arm I (Nivolumab, Gemcitabine, Cisplatin / Carboplatin) | Arm II (Gemcitabine, Cisplatin / Carboplatin)
Number analyzed (Participants) | 8 | 3
score on a scale | 63.9 (9.6) | 75.0 (4.8)

10. Secondary Outcome: Multidimensional Fatigue Inventory (MFI)-20 Total Score
Description: The MFI-20 is a 20-item self-report instrument measuring fatigue with the total score ranging from 20 to 100 and a higher score indicating more fatigue.
Time Frame: End of cycle 6 (each cycle is 21 days)
Population: Randomized participants with MFI data at cycle 6
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Arm I (Nivolumab, Gemcitabine, Cisplatin / Carboplatin) | Arm II (Gemcitabine, Cisplatin / Carboplatin)
Number analyzed (Participants) | 8 | 3
score on a scale | 61.6 (4.4) | 72.7 (7.8)

11. Secondary Outcome: Progression-free Survival by Programmed Death Receptor Ligand-1 (PD-L1) Combined Positive Score (CPS) and Tumor Proportion Score (TPS)
Description: This study hypothesizes that the use of PD-L1 expression based on the TPS or CPS may be useful in identifying those patients who are more likely to benefit from treatment with PD-1 inhibitor in combination with chemotherapy. This study will explore a range of CPS and TPS scores.
Time Frame: Baseline to the date of failure or last known follow-up. Maximum follow-up time was 2.3 years.
Population: No assays were performed, and no data were collected for this outcome measure.
Arm/Group | Arm I (Nivolumab, Gemcitabine, Cisplatin / Carboplatin) | Arm II (Gemcitabine, Cisplatin / Carboplatin)
Number analyzed (Participants) | 0 | 0

12. Other Pre Specified Outcome: Overall Survival by PD-L1 CPS and TPS
Description: as for outcome 11
Time Frame: Baseline to the date of failure or last known follow-up. Maximum follow-up time was 2.3 years.
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Change From Baseline to Cycle 6 in Global Heath Status (GHS) Score of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30)
Description: Global Health Status is calculated from two questions on the EORTC QLQ-C30. The question responses range from 1 "very poor" to 7 "excellent" such that a higher response indicates better quality of life (QOL). The mean of these responses is linearly transformed to a range of 0 (worst) to 100 (best). Change is calculated as later value minus baseline value such that a positive change indicates improvement
Time Frame: Baseline and end of cycle 6 (each cycle is 21 days)
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Change From Baseline to Cycle 6 in Multidimensional Fatigue Inventory (MFI)-20 Total Score
Description: The MFI-20 is a 20-item self-report instrument measuring fatigue with the total score ranging from 20 to 100 and a higher score indicating more fatigue. Change is calculated as later value minus baseline value such that a negative change indicates decreased fatigue.
Time Frame: Baseline and end of cycle 6 (each cycle is 21 days)
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Translational Research Studies
Time Frame: From randomization to last follow-up, assessed up to 8 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Baseline to the date of failure or last known follow-up. Maximum follow-up time was 2.3 years.
Groups:
- Arm I (Nivolumab, Gemcitabine, Cisplatin / Carboplatin): Six cycles (3 weeks each):
  * Nivolumab 360 mg fixed dose IV over 30 minutes on day 1.
  * Cisplatin 80 mg/m^2 IV over 30-60 minutes or carboplatin AUC of 5 on day 1.
  * Gemcitabine 1000 mg/m^2 in IV over 30 minutes on days 1 and 8.
  Followed by maintenance therapy for up to 24 cycles (4 weeks each):
  * Nivolumab 480 mg fixed dose IV over 30 minutes on day 1.
Arm/Group | Arm I (Nivolumab, Gemcitabine, Cisplatin / Carboplatin) | Arm II (Gemcitabine, Cisplatin / Carboplatin)
All-Cause Mortality (participants affected / at risk) | 3/11 | 0/4
Serious Adverse Events (participants affected / at risk) | 10/11 | 2/4
Other Adverse Events (participants affected / at risk) | 11/11 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Nivolumab, Gemcitabine, Cisplatin / Carboplatin) (N=11) | Arm II (Gemcitabine, Cisplatin / Carboplatin) (N=4)
Anemia (Blood and lymphatic system disorders) | 5 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1
Alkaline phosphatase increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 6 | 2
Platelet count decreased (Investigations) | 1 | 0
White blood cell decreased (Investigations) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Nivolumab, Gemcitabine, Cisplatin / Carboplatin) (N=11) | Arm II (Gemcitabine, Cisplatin / Carboplatin) (N=4)
Anemia (Blood and lymphatic system disorders) | 5 | 2
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 | 2
Hearing impaired (Ear and labyrinth disorders) | 2 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Hypophysitis (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 2 | 0
Dry eye (Eye disorders) | 1 | 0
Eye disorders - Other (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 6 | 3
Diarrhea (Gastrointestinal disorders) | 0 | 2
Dry mouth (Gastrointestinal disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 3
Dysphagia (Gastrointestinal disorders) | 4 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 2 | 3
Nausea (Gastrointestinal disorders) | 5 | 3
Oral hemorrhage (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2
Chills (General disorders) | 1 | 1
Edema limbs (General disorders) | 2 | 1
Fatigue (General disorders) | 7 | 3
Fever (General disorders) | 3 | 0
General disorders and administration site conditions - Other (General disorders) | 1 | 0
Localized edema (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Allergic reaction (Immune system disorders) | 0 | 1
Infections and infestations - Other (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Mucosal infection (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Thrush (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 2
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 2
Alkaline phosphatase increased (Investigations) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 2
Blood bicarbonate decreased (Investigations) | 1 | 0
Creatinine increased (Investigations) | 2 | 1
Investigations - Other (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 7 | 3
Platelet count decreased (Investigations) | 3 | 2
Weight loss (Investigations) | 3 | 1
White blood cell decreased (Investigations) | 3 | 2
Anorexia (Metabolism and nutrition disorders) | 4 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 3 | 0
Hyponatremia (Metabolism and nutrition disorders) | 3 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Concentration impairment (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 1
Dysgeusia (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 2 | 2
Lethargy (Nervous system disorders) | 1 | 0
Nystagmus (Nervous system disorders) | 1 | 0
Paresthesia (Nervous system disorders) | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 1
Syncope (Nervous system disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 5 | 1
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 0
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Flushing (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Superficial thrombophlebitis (Vascular disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
This study stopped accrual early at 15 participants of the 316 planned, due to published results of two other studies resolving the study question (NCT03707509, NCT03581786). As less than 5% of the sample size was accrued, no statistical testing was done.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-16): https://cdn.clinicaltrials.gov/large-docs/09/NCT04458909/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-16): https://cdn.clinicaltrials.gov/large-docs/09/NCT04458909/ICF_001.pdf